CLINICAL TRIAL: NCT01285960
Title: A Clinical Study to Evaluate Safety of the ExAblate Model 2100 Type 1.1 System (ExAblate 2100/2000 UF V2 System) in the Treatment of Symptomatic Uterine Fibroids
Brief Title: ExAblate UF V2 System for the Treatment of Symptomatic Uterine Fibroids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UF031
Record Dates: First submitted 2011-01-27; First posted 2011-01-28 (Estimated); Results first posted 2019-02-19 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-02

CONDITIONS: Uterine Fibroids
Keywords: Uterine fibroids; MRgFUS; ExAblate; Focused Ultrasound; Symptomatic uterine fibroids
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ExAblate treatment UF V2 (Experimental): ExAblate MRgFUS Treatment
  Interventions: Device: ExAblate Treatment UF V2

INTERVENTIONS:
Device: ExAblate Treatment UF V2 — Treatment with the ExAblate UF V2 system. Patients may have up to two ExAblate treatments within a two-week period.

SUMMARY:
The purpose of this study is to evaluate the safety and ablation efficacy of the ExAblate UF V2 System when treating symptomatic uterine fibroids.

The ExAblate System is a medical device that involves a focused ultrasound system and an MRI scanner. ExAblate delivers a pulse of focused ultrasound energy, or sonication, to the targeted tissue. In this particular study, the targeted tissue is uterine fibroids. Each sonication is used to heat small spots in the fibroid much like a magnifying glass can be used to focus light to heat a spot. The heat created kills a portion of the fibroid with the goal of decreasing or eliminating uterine fibroid-related symptoms. Repeated sonications are performed until the entire fibroid is treated or the treated volume is determined to be appropriate.

The ExAblate system is commercially approved in the United States to treat symptomatic uterine fibroids.

The ExAblate UF V2 System is an experimental device and is being investigated in this study. While similar to the commercial system, the ExAblate UF V2 device includes the following major changes, among others, which are intended to improve device performance and safety:

* Up and down movement of the ultrasound transducer, in an attempt to improve fibroid treatment by moving the ultrasound focal point within the targeted fibroid.
* Ultrasound energy can be turned off for a specific area in an attempt to minimize amount of energy passing through sensitive areas of the body.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age 18 or older
2. Patients who present with symptomatic uterine fibroids and are not seeking treatment for the reason of improving fertility.
3. Patients who have given written informed consent
4. Patients who are able and willing to attend all study visits
5. Patients who are pre or peri-menopausal (within 12 months of last menstrual period)
6. Patients should have completed child bearing
7. Able to communicate sensations during the ExAblate procedure.
8. Uterine fibroids, which are device accessible (i.e., positioned in the uterus such that they can be accessed without being shielded by bowel or bone).
9. Fibroid(s) clearly visible on non-contrast MRI.

Exclusion Criteria:

1. Pregnant patients, as confirmed by serum/urine test at time of screening, or urine pregnancy test on the day of treatment. Pregnancies following ExAblate treatment could be dangerous for both mother and fetus.
2. Uterine size >24 weeks.
3. Patients with pedunculated fibroids
4. Patients with active pelvic inflammatory disease (PID).
5. Patients with active local or systemic infection
6. Patients experiencing any symptoms of lower extremity neuropathy, including chronic leg or lower back pain, within the last 6 months
7. Contraindication for MRI Scan:

   * Severe claustrophobia that would prevent completion of procedure in the MR unit
   * Metallic implants that are incompatible with MRI
   * Sensitivity to MRI contrast agents
   * Any other contraindication for MRI Scan
8. Extensive abdominal scarring in the beam path (that cannot be avoided by redirection of the beam)
9. Dermoid cyst of the ovary anywhere in the treatment path.
10. Known or suspected pelvic carcinoma or pre-malignant conditions, including sarcoma and adenomatous hyperplasia.
11. Intrauterine device (IUD) anywhere in the treatment path
12. Undiagnosed vaginal bleeding

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2012-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Duke University, Durham, North Carolina
  - Ohio Health Research Institute, Columbus, Ohio
  - University of Virginia Health System, Charlottesville, Virginia

REFERENCES:
- [Derived] Bitton RR, Fast A, Vu KN, Lum DA, Chen B, Hesley GK, Raman SS, Matsumoto AH, Price TM, Tempany C, Dhawan N, Dolen E, Kohi M, Fennessey FM, Ghanouni P. What predicts durable symptom relief of uterine fibroids treated with MRI-guided focused ultrasound? A multicenter trial in 8 academic centers. Eur Radiol. 2023 Nov;33(11):7360-7370. doi: 10.1007/s00330-023-09984-4. Epub 2023 Aug 9. PMID 37553488
- See also: Sponsor's Web Page — https://www.insightec.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ExAblate Treatment UF V2
Started | 108 (2 subjects receiving fewer than 10 sonications were added to the 106 for safety population of 108)
Completed | 102 (An additional 2 subjects receiving fewer than 10 sonications were included in the safety population)
Not Completed | 6
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 2
Not completed — 2 subjects received less 10 sonications | 2

BASELINE CHARACTERISTICS:
Population: 106 subjects received the ExAblate UF V2 treatment. Two (2) additional subjects receiving fewer than 10 sonications were included in the safety sample (108 subjects)
Arm/Group | ExAblate Treatment UF V2
Number analyzed (Participants) | 108
Age, Continuous [Mean (Full Range); unit: years] | 46 [31 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108
  Male | 0
Race/Ethnicity, Customized [Number; unit: %]
  European/Middle East (White) | 69
  African American | 14
  Asian | 13
  Hispanic | 5
Region of Enrollment [Number; unit: participants]
  United States | 108

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Leg Pain or Lower Extremity Neuropathy Persisting or Occuring Greater Than 10 Days Following Treatment
Description: The hypothesis for this study was that the percentage of subjects experiencing persistent leg pain would be less than 10%
Time Frame: From treatment to 1-month post-treatment
Population: Per protocol 2 subjects receiving < 10 sonications were excluded from the safety sample size of 108 for an primary safety analysis sample size of 106.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ExAblate Treatment UF V2
Number analyzed (Participants) | 106
Percentage of participants | 0 [0 to 5.6]

ADVERSE EVENTS:
Time Frame: 1 month
Description: 2 subjects receiving fewer than 10 sonications were added to the sample size of 106 treated subjects for a total safety sample size of 108
Arm/Group | ExAblate Treatment UF V2
All-Cause Mortality (participants affected / at risk) | 0/108
Serious Adverse Events (participants affected / at risk) | 1/108
Other Adverse Events (participants affected / at risk) | 102/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ExAblate Treatment UF V2 (N=108)
Acute Bowel Perforation (Gastrointestinal disorders) | 1 (1) — Device-Treatment Related AE
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ExAblate Treatment UF V2 (N=108)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Skin burn (Skin and subcutaneous tissue disorders) | 3 (3)
Itching (Skin and subcutaneous tissue disorders) | 1 (1)
Small bruise at IV Site (Skin and subcutaneous tissue disorders) | 1 (1)
Edema/Hypo-intense tissu (Surgical and medical procedures) | 7 (10)
Nausea/vomiting (Surgical and medical procedures) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Nausea/vomiting (Gastrointestinal disorders) | 2 (4)
Generalized GI upset and decreased activity (Gastrointestinal disorders) | 1 (1)
Stomach cramping (Gastrointestinal disorders) | 1 (1)
Bloody mucus in stool (Gastrointestinal disorders) | 1 (1)
Abdominal cramping (Reproductive system and breast disorders) | 2 (2)
Dyspareunia (Reproductive system and breast disorders) | 1 (1)
Menstrual cramping (Reproductive system and breast disorders) | 1 (1)
Back pain during period (Reproductive system and breast disorders) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1)
Vaginal bleeding between periods (Reproductive system and breast disorders) | 4 (4)
Anxiety (Psychiatric disorders) | 1 (1)
Leg/calf pain (Nervous system disorders) | 2 (2)
Dizziness/vertigo (Nervous system disorders) | 2 (2)
Tingling sensation in spine (Nervous system disorders) | 1 (1)
Left leg anterior compartment tenderness (General disorders) | 1 (1)
Decreased sensation in right foot (General disorders) | 1 (1)
IV infiltration (General disorders) | 1 (1)
Position Pain (Surgical and medical procedures) | 23 (23)
Sonication Pain (Surgical and medical procedures) | 55 (73)
Sonication-related epidermal pain (Surgical and medical procedures) | 49 (57)
Sonication related neuromuscular pain (Surgical and medical procedures) | 81 (121)
Fatigue (General disorders) | 2 (2)
Fever/chills (Surgical and medical procedures) | 4 (5)
Post-embolization like symptoms (Blood and lymphatic system disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 4 (4)
Increased urinary frequency (Renal and urinary disorders) | 1 (1)
Pain or burning at urinary catheter site (Renal and urinary disorders) | 2 (2)
Difficulty initiating urination (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary tract infection (UTI) (Renal and urinary disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No